CLINICAL TRIAL: NCT07394400
Title: A Comprehensive Assessment of the Impact of Gender-Affirming Hormone Therapy on Cardiovascular Risk, Metabolic Health, and Mood Disorders in Transgender Individuals.
Brief Title: Effects of Gender-Affirming Hormone Therapy on Cardiovascular, Metabolic, and Mental Health Outcomes in Transgender Adults.
Status: Not yet recruiting | Type: Observational
Sponsor: Milagros Rocha Barajas (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Milagros Rocha Barajas, Senior Postdoctoral Researcher, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: PI25/01841
Record Dates: First submitted 2026-01-13; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Transgender Individuals
Keywords: GAHT; inflammation; atherosclerosis; periodontal disease; Transgender
MeSH Terms: conditions — Inflammation; Atherosclerosis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Serum, neutrophils and Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to examine the impact of gender-affirming hormone therapy (GAHT) on mood in transgender individuals and to explore its potential association with early atherosclerotic processes. The main questions it aims to answer are:

* Whether GAHT in transgender individuals has a psychological and functional impact, assessed through mood, stress, and self-esteem. Additionally, the study will analyze whether morphofunctional changes (including body composition, muscle strength, cardiorespiratory fitness, and metabolic flexibility) are related to inflammatory responses and psychological well-being.
* Whether the administration of GAHT poses a cardiovascular risk by influencing biochemical, inflammatory, and oxidative markers, mitochondrial function, and the activation of the NLRP3 inflammasome in leukocytes.

Participants will undergo evaluation of early stages of the atherosclerotic process through the analysis of leukocyte-endothelial interactions, adhesion molecule expression, and ankle-brachial index (ABI), as well as periodontal parameters. Overall, this study aims to contribute to improving healthcare delivery and promoting more equitable and gender-affirming medical services tailored to the needs of transgender individuals.

DETAILED DESCRIPTION:
Blood samples will be collected from patients at baseline (before starting gender-affirming hormone therapy), 6 and 12 months after. From fasting blood samples (12h), peripheral blood mononuclear cells (PBMCs) and neutrophil fractions will be isolated using an immunomagnetic method, following the manufacturer's protocol, and plasma and serum will be stored at -80°C until analysis. LUNA-FL will be used to determine cell count and viability (acridine orange and propidium iodide double stain) in cell samples.

For periodontal assessment participants will undergo a comprehensive periodontal examination to determine several gingival parameters, including probing depth (PD), clinical attachment loss (CAL), bleeding index, plaque index, and calculus. Based on these data, the presence or absence of periodontal disease, as well as its extent when present, will be diagnosed.

Biochemical parameters of carbohydrate metabolism - glucose, insulin, glycated hemoglobin (A1c) -, lipid profile - total cholesterol, LDL, HDL, triglycerides (TG), apolipoproteins AI and B -, emerging inflammatory and cardiovascular risk markers - C-Reactive Protein (CRP), C3c, and retinol-binding protein 4 (RBP4) -, and complete blood count will be determined at the hospital's Clinical Analysis Service. Weight, height, and blood pressure will be measured using standardized methods.

Morphofunctional changes will be assessed at baseline and after 12 months of GAHT. Participants will attend the Morphofunctional Assessment Unit after an overnight fast. Body composition and hydration status will be measured using bioelectrical impedance analysis (mBCA 520, SECA, Germany). The quality and distribution of adipose and muscle tissue will be evaluated through Nutritional Ultrasound® using a DP-50 Expert Mobile Ultrasound System (Mindray®) equipped with a multifrequency linear transducer (5-10 MHz). Measurements will be performed in B-mode following established methodological recommendations (10.1016/j.endinu.2022.03.008).

For evaluation of cardiorrespiratory fitness through an incremental ramp exercise test on a cycle ergometer (Ergoselect 200 P, Ergoline, Germany) performed to voluntary exhaustion, following established recommendations (10.1152/ajpregu.00126.2020.0363-6119/20), to determine VO₂max and ventilatory thresholds. A COSMED K5 metabolic analyzer (COSMED, Italy) will be used for gas exchange analysis. Blood pressure, heart rate (Polar H10 heart rate monitor; Polar Electro Oy, Finland), and oxygen saturation at both systemic and muscular levels (WristOx2 3150, Nonin Medical Inc., USA; and Moxy®, Fortiori Design LLC, USA, respectively) will be continuously monitored. Maximal isometric strength of the knee extensor muscles will be measured using a MicroFET2 dynamometer (Hoggan Scientific LLC, USA), and resting metabolic rate (RMR) will also be assessed with the COSMED K5 metabolic analyzer.

For detection of differences in protein expression, cells will be incubated in lysis buffer with protease and phosphatase inhibitors (RIPA Buffer) for 15 minutes at 4 degrees celsius (°C). The supernatant will be collected after centrifugation for 15 minutes at 16,000g. The total protein concentration will be quantified using a bicinchoninic acid (BCA) protein assay. Aliquots of 25 µg of protein will be resolved on 8-16% gradient SDS-polyacrylamide gels and transferred to nitrocellulose membranes. Target proteins will be detected by incubating the membranes with anti-actin, JNK, NFkB, NLRP3, ASC, caspase 1, NADPH oxidase, catalase, GPX1, SOD1, NRF2, mitochondrial markers such as the different complexes of the electron transport chain and PGC1α. The protein signal will be detected by chemiluminescence and analyzed by densitometry.

To measure the expression of the anti-oxidant enzymes SOD1, NFR2 and the genes dependent on the NRF2 antioxidant pathway (such as GPX1, GCLC, GLCM and TXNRD1) using real-time PCR. Mitochondrial function will be assessed by analysing PBMC oxygen consumption using the Seahorse XF technique (Agilent) as described in 10.1016/j.redox.2025.103516.

Inflammasome activation in PBMCs will be evaluated by detecting ASC specks using fluorescence microscopy. Briefly, PBMCs will be seeded on coverslips coated with Poly-D-Lysine, fixed with paraformaldehyde (PFA) 4% for 20 minutes, permeabilized with Triton X-100 for 20 minutes and blocking with Phosphate-buffered saline buffer-Bovine serum albumn (PBS-BSA) 3% for 1 hour at room temperature. Hybridization with specific primary antibodies (diluted in PBS-BSA 1%) will be carry out overnight at 4 ºC and then, secondary antibodies conjugated with AlexaFluor fluorophores will be incubated for 1 hour in the dark at room temperature. Stained samples will be transferred the coverslip onto microscope slide and conserved in anti-fade fluorescence mounting medium.

Gene expression profiling will be performed using the Nanostring® nCounter® platform to identify transcripts differentially expressed after 12 months of THAG intervention. The multiplex metabolism panel, encompassing 768 genes, will target pathways involved in inflammation (TLR, NF-κB), oxidative stress, cytokine signaling, and mitochondrial respiration. Data analysis will be conducted using the nSolver software (Nanostring Technologies). All experiments will be outsourced to Diagnostica Longwood, S.L.

Circulating levels of cytokines, adhesion molecules and serum oxidative stress markers will be measured in serum samples. This samples will be analyzed with a Luminex® 200 analyzer system following the Milliplex® MAP Kit manufacturer's procedure.

A parallel plate flow chamber, connected to an inverted microscope, will enable the researchers to measure neutrophil-endothelial cell interactions in vitro. Through this system, the leukocyte suspension obtained from patients will be perfused over a monolayer of immortalized endothelial cells (HUVEC/TERT 2) under conditions simulating blood flow. Videos will be analyzed afterward to determine flow, rolling velocity, and firm adhesion of leukocytes to endothelial cells, as previously described (Antioxidants. 2020 Aug 11;9(8):734).

DNA will also be extracted from serum according to the "blood and body fluid protocol" of the QIAamp blood reagent set (QIAgen, Hilden, Germany); 200 μL of plasma will be applied to each column, DNA will be eluted in 100 μL of supplied buffer and will be stored at -20°C until use. mtDNA will be quantified with reverse transcription-quantitative polymerase chain reaction (RT-qPCR) using specific primers for obtaining circulating mtDNA levels.

Data analysis will be performed with SPSS 17.0. Groups will be compared using unpaired Student's t-tests or Mann-Whitney U tests for parametric and non-parametric data, respectively. Changes after intervention will be evaluated using paired Student's t-tests or Wilcoxon tests, depending on the variable distribution. Pearson or Spearman correlation coefficients will be used to measure the strength of association between variables. In multivariable regression models, the relationship between two or more explanatory variables (independent variables) and a response variable (dependent variable) will be evaluated by fitting a linear equation to the obtained data. Qualitative data will be expressed in percentages, and proportions will be compared using a Chi-square test. All tests will use a 95% confidence interval, and differences will be considered statistically significant when p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Trans men and trans women over the age of 16

Exclusion Criteria:

* systemic inflammatory diseases
* uncontrolled infections
* severe autoimmune diseases intersex biological conditions (resistance, severe sexual development or chromosomal abnormalities, congenital adrenal hyperplasia)
* treatment with metformin, statins or oral contraceptives in the previous 6 months
* serious life-threatening diseases
* diseases that compromise follow-up
* BMI higher than 35

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Transgender individuals referred to a Gender Identity Unit who are requesting Gender Affirmation Hormone Therapy for the first time. It will consist of three visits: at the start, and after 6 and 12 months of treatment.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the degree of activation of the inflammasome complex in transgender individuals following gender-affirming hormone therapy. | At recruitment
  Relative protein expression of NLRP3, ASC, Caspase-1 and inflammatory mediators NFκB, JNK by Western Blot and normalized to the loading control protein in PBMC. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in endothelial function in the study population. | At recruitment
  Evaluation of leucocytes adhesion to the endothelial cell in vitro by means of a parallel flow chamber system coupled to an inverted phase-contrast microscope. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in endothelial function at molecular level in the study population. | At recruitment
  Evaluation of circulating levels of adhesion molecules - P-selectin, ICAM-1, and VCAM-1, levels of the pro-oxidant enzyme MPO and circulating cytokines (L1β, IL18, IL6, IL10 and TNFα) in serum using Luminex technique. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in the systemic inflammation status in the study population. | At recruitment
  Evaluation of circulating levels of mtDNA in serum samples using RT-PCR. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in the expression of genes related to inflammatory pathways in PBMC in the study population. | At recruitment
  Identification of altered messengers using a metabolic multiplex panel, evaluating genes of interest in inflammatory pathways (TLR and NFkB), oxidative stress, cytokine signalling, and mitochondrial respiration. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in the expression of genes related to oxidative stress levels in PBMC in the study population. | At recruitment
  Relative expression of genes related to oxidative stress (SOD1, NRF2, GSR, GPX1, GCLC, GCLM and TXNRD1) by PCR real time. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in the expression of genes related to cellular respiration in PBMC in the study population. | At recruitment
  Relative expression of pro and antioxidants enzimes (NADPH oxidase, catalase, GPX1, SOD1, and NFR2) and genes related to mitochondrial respiration (I, II, III, IV and V complexes) and PGC1α in PBMC by WB. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Changes in the degree of activation of the inflammasome complex in transgender individuals following gender-affirming hormone therapy. | At recruitment
  Study of inflammasome assembly by confocal microscopy in PBMC. This measurement will be taken at the start, and at 6 and 12 months of THAG.

SECONDARY OUTCOMES:
Evaluation of redox status (PBMCs and PMNs) in the study population. | At recruitment
  Determination of redox status using flow cytometry with fluorescent probes. This measurement will be taken at the start, and at 6 and 12 months of THAG.
Evaluation of mitochondrial function of leukocytes (PBMCs and PMNs) in the study population. | At recruitment
  Determination of mitochondrial function by analysing oxygen consumption in PBMCs using the Seahorse XF technique (Agilent). This measurement will be taken at the start, and at 6 and 12 months of THAG.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rocha, PhD, Principal Investigator — FISABIO-HOSPITAL DR PESET
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Valencia, Spain

REFERENCES:
- [Background] Koukoulis GN, Filiponi M, Gougoura S, Befani C, Liakos P, Bargiota Alpha. Testosterone and dihydrotestosterone modulate the redox homeostasis of endothelium. Cell Biol Int. 2022 Apr;46(4):660-670. doi: 10.1002/cbin.11768. Epub 2022 Jan 30. PMID 35066972
- [Background] Exposito-Campos P, Gomez-Balaguer M, Hurtado-Murillo F, Morillas-Arino C. Evolution and trends in referrals to a specialist gender identity unit in Spain over 10 years (2012-2021). J Sex Med. 2023 Feb 27;20(3):377-387. doi: 10.1093/jsxmed/qdac034. PMID 36763946
- [Background] Banuls C, Rovira-Llopis S, Martinez de Maranon A, Veses S, Jover A, Gomez M, Rocha M, Hernandez-Mijares A, Victor VM. Metabolic syndrome enhances endoplasmic reticulum, oxidative stress and leukocyte-endothelium interactions in PCOS. Metabolism. 2017 Jun;71:153-162. doi: 10.1016/j.metabol.2017.02.012. Epub 2017 Feb 27. PMID 28521868
- [Background] Zhang Q, Goodman M, Adams N, Corneil T, Hashemi L, Kreukels B, Motmans J, Snyder R, Coleman E. Epidemiological considerations in transgender health: A systematic review with focus on higher quality data. Int J Transgend Health. 2020 Apr 15;21(2):125-137. doi: 10.1080/26895269.2020.1753136. eCollection 2020. PMID 33015664
- [Background] Victor VM, Rovira-Llopis S, Banuls C, Diaz-Morales N, Castello R, Falcon R, Gomez M, Rocha M, Hernandez-Mijares A. Effects of metformin on mitochondrial function of leukocytes from polycystic ovary syndrome patients with insulin resistance. Eur J Endocrinol. 2015 Nov;173(5):683-91. doi: 10.1530/EJE-15-0572. Epub 2015 Aug 28. PMID 26320144
- [Background] Villar CC, Sloniak MC, de Assis JB, Porto RC, Romito GA. Unveiling sex-disparities and the impact of gender-affirming hormone therapy on periodontal health. Front Dent Med. 2024 Sep 16;5:1430193. doi: 10.3389/fdmed.2024.1430193. eCollection 2024. PMID 39917660
- [Background] Nokoff NJ, Nemkov T, Bothwell S, Cree MG, Fuller KNZ, Keller AC, Kelsey MM, Nadeau KJ, Moreau KL. Differences in cardiorespiratory fitness by gonadotropin-releasing hormone agonist treatment before and after testosterone in transgender adolescents. J Appl Physiol (1985). 2024 Nov 1;137(5):1470-1483. doi: 10.1152/japplphysiol.00629.2024. Epub 2024 Oct 17. PMID 39417821
- [Background] Cheung AS, Zwickl S, Miller K, Nolan BJ, Wong AFQ, Jones P, Eynon N. The Impact of Gender-Affirming Hormone Therapy on Physical Performance. J Clin Endocrinol Metab. 2024 Jan 18;109(2):e455-e465. doi: 10.1210/clinem/dgad414. PMID 37437247
- [Background] Lakshmikanth T, Consiglio C, Sardh F, Forlin R, Wang J, Tan Z, Barcenilla H, Rodriguez L, Sugrue J, Noori P, Ivanchenko M, Pinero Paez L, Gonzalez L, Habimana Mugabo C, Johnsson A, Ryberg H, Hallgren A, Pou C, Chen Y, Mikes J, James A, Dahlqvist P, Wahlberg J, Hagelin A, Holmberg M, Degerblad M, Isaksson M, Duffy D, Kampe O, Landegren N, Brodin P. Immune system adaptation during gender-affirming testosterone treatment. Nature. 2024 Sep;633(8028):155-164. doi: 10.1038/s41586-024-07789-z. Epub 2024 Sep 4. PMID 39232147
- [Background] Glintborg D, Christensen LL, Andersen MS. Transgender healthcare: metabolic outcomes and cardiovascular risk. Diabetologia. 2024 Nov;67(11):2393-2403. doi: 10.1007/s00125-024-06212-6. Epub 2024 Jul 3. PMID 38958699
- [Background] Coleman E, Radix AE, Bouman WP, Brown GR, de Vries ALC, Deutsch MB, Ettner R, Fraser L, Goodman M, Green J, Hancock AB, Johnson TW, Karasic DH, Knudson GA, Leibowitz SF, Meyer-Bahlburg HFL, Monstrey SJ, Motmans J, Nahata L, Nieder TO, Reisner SL, Richards C, Schechter LS, Tangpricha V, Tishelman AC, Van Trotsenburg MAA, Winter S, Ducheny K, Adams NJ, Adrian TM, Allen LR, Azul D, Bagga H, Basar K, Bathory DS, Belinky JJ, Berg DR, Berli JU, Bluebond-Langner RO, Bouman MB, Bowers ML, Brassard PJ, Byrne J, Capitan L, Cargill CJ, Carswell JM, Chang SC, Chelvakumar G, Corneil T, Dalke KB, De Cuypere G, de Vries E, Den Heijer M, Devor AH, Dhejne C, D'Marco A, Edmiston EK, Edwards-Leeper L, Ehrbar R, Ehrensaft D, Eisfeld J, Elaut E, Erickson-Schroth L, Feldman JL, Fisher AD, Garcia MM, Gijs L, Green SE, Hall BP, Hardy TLD, Irwig MS, Jacobs LA, Janssen AC, Johnson K, Klink DT, Kreukels BPC, Kuper LE, Kvach EJ, Malouf MA, Massey R, Mazur T, McLachlan C, Morrison SD, Mosser SW, Neira PM, Nygren U, Oates JM, Obedin-Maliver J, Pagkalos G, Patton J, Phanuphak N, Rachlin K, Reed T, Rider GN, Ristori J, Robbins-Cherry S, Roberts SA, Rodriguez-Wallberg KA, Rosenthal SM, Sabir K, Safer JD, Scheim AI, Seal LJ, Sehoole TJ, Spencer K, St Amand C, Steensma TD, Strang JF, Taylor GB, Tilleman K, T'Sjoen GG, Vala LN, Van Mello NM, Veale JF, Vencill JA, Vincent B, Wesp LM, West MA, Arcelus J. Standards of Care for the Health of Transgender and Gender Diverse People, Version 8. Int J Transgend Health. 2022 Sep 6;23(Suppl 1):S1-S259. doi: 10.1080/26895269.2022.2100644. eCollection 2022. PMID 36238954